CLINICAL TRIAL: NCT03528343
Title: Comparing Narcotic vs. Non-narcotic Pain Regimens After Pediatric Appendectomy: A Randomized Controlled Trial
Brief Title: Narcotic vs. Non-narcotic Pain Regimens After Pediatric Appendectomy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lost research support for enrolling patients
Sponsor: University of Utah (Other)
Collaborators: Primary Children's Hospital (Other)
Responsible Party: Principal Investigator, Sean Stokes, General Surgery Resident, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU83426
Record Dates: First submitted 2017-09-12; First posted 2018-05-17 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Appendicitis; Pain, Postoperative
Keywords: appendicitis; postoperative pain; patient satisfaction; children; pediatric; narcotic; pain control
MeSH Terms: conditions — Appendicitis; Pain, Postoperative; Patient Satisfaction; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tylenol/Motrin (Experimental): Group of patients who will receive instructions to use tylenol and motrin for pain control, and parents will be sent home with a paper prescription with a rescue does of standard of care narcotics. They will be instructed to only use the rescue dose if pain is uncontrolled using over the counter medications.
  Interventions: Drug: Non-narcotic pain control
- Narcotic (No Intervention): Group of patients who will receive the standard of care narcotic prescription filled upon discharge.

INTERVENTIONS:
Drug: Non-narcotic pain control — Education to use tylenol and motrin only for pain control unless this is unable to control pain. Rescue prescription provided.
  Arms: Tylenol/Motrin

SUMMARY:
There is concern that pain prescription after outpatient pediatric surgical procedures is excessive and is in excess of patient need. Current practice following pediatric appendectomy is to prescribe all children with 5-15 doses of narcotic pain medication upon discharge regardless of their age, severity of appendicitis, or pain control in the hospital. This study examines the amount of narcotic pain control required by pediatric patients after undergoing appendectomy using a randomized controlled trial study design.

Pain control will be assessed with a post-operative pain scale, patient satisfaction survey, and parent satisfaction survey on the days following surgery and at post-operative follow-up.

The hypothesis is that the pain scores and patient satisfaction surveys will show no difference in post-operative pain control between the two arms.

DETAILED DESCRIPTION:
There is concern that pain prescription after outpatient pediatric surgical procedures is excessive and is in excess of patient need. Current practice following pediatric appendectomy is to prescribe all children with 5-15 doses of narcotic pain medication upon discharge regardless of their age, severity of appendicitis, or pain control in the hospital. This study examines the amount of narcotic pain control required by pediatric patients after undergoing appendectomy using a randomized controlled trial study design.

Children admitted after undergoing surgical management for a diagnosis of acute appendicitis will be randomized at discharge to a narcotic arm or a tylenol/motrin arm. The narcotic arm will receive the standard of care narcotic prescription. The tylenol/motrin arm will receive education to use tylenol and motrin for pain control as well as a paper prescription provided for the sole purpose of rescue.

Pain control will be assessed with a post-operative pain scale, patient satisfaction survey, and parent satisfaction survey on the days following surgery and at post-operative follow-up.

The hypothesis is that the pain scores and patient satisfaction surveys will show no difference in post-operative pain control between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0 to 18 years old
* Patients have undergone appendectomy by any technique (open, laparoscopic, single-port)

Exclusion Criteria:

* Patients on chronic opioids
* Patient undergoes a more extensive or additional procedures at the time of operation due to complications or other indication
* Pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Parental pain control satisfaction using Parental Post-operative Pain Measure (PPPM) | 2-week follow-up visit
  Parental satisfaction with pain control at home following pediatric appendectomy as assessed by the validated Parental Post-operative Pain Measure (PPPM)

SECONDARY OUTCOMES:
Parental pain control satisfaction using Parental Post-operative Pain Measure (PPPM) | Changes from in-hospital, days 1-3 following discharge, and 2-week follow-up
  Parental satisfaction with pain control at home following pediatric appendectomy as assessed by Parental Post-operative Pain Measure (PPPM)
Patient pain control satisfaction using adaptation of Parental Post-operative Pain Measure (PPPM) | Changes from in-hospital, days 1-3 following discharge, and 2-week follow-up
  Patient satisfaction with pain control at home following pediatric appendectomy as assessed by an adaptation of Parental Post-operative Pain Measure (PPPM)
Patient pain scores using Wong-Baker Faces Pain Rating Scale | Changes from in-hospital, days 1-3 following discharge, and 2-week follow-up
  Patient description of pain control using validated Wong-Baker Faces Pain Rating Scale. This scale presents the subject with a series of 6 depictions of faces and a text description of pain level. The range is from 0 "No Hurt" to 10 "Hurts Worst".
Number of pain medications used | Post-operative days 1-14 (until follow-up)
  Number of pain medications used
Days of pain medication requirement after discharge | Post-operative days 1-14 (until follow-up)
  Number of days patient required pain medication
Number of pain medication side effects | Post-operative days 1-14 (until follow-up)
  Side effects experienced by taking pain medications following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Fenton, MD, Principal Investigator — University of Utah, Primary Children's Hospital
Locations (1):
- Primary Children's Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blakely ML, Spurbeck WW, Lobe TE. Current status of laparoscopic appendectomy in children. Semin Pediatr Surg. 1998 Nov;7(4):225-7. doi: 10.1016/s1055-8586(98)70035-6. PMID 9840903
- [Background] Buckius MT, McGrath B, Monk J, Grim R, Bell T, Ahuja V. Changing epidemiology of acute appendicitis in the United States: study period 1993-2008. J Surg Res. 2012 Jun 15;175(2):185-90. doi: 10.1016/j.jss.2011.07.017. Epub 2011 Aug 9. PMID 22099604
- [Background] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Background] Alkhoury F, Knight C, Stylianos S, Zerpa J, Pasaron R, Mora J, Aserlind A, Malvezzi L, Burnweit C. Prospective Comparison of Nonnarcotic versus Narcotic Outpatient Oral Analgesic Use after Laparoscopic Appendectomy and Early Discharge. Minim Invasive Surg. 2014;2014:509632. doi: 10.1155/2014/509632. Epub 2014 Apr 14. PMID 24834350
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704
- [Background] Abou-Karam M, Dube S, Kvann HS, Mollica C, Racine D, Bussieres JF, Lebel D, Nguyen C, Thibault M. Parental Report of Morphine Use at Home after Pediatric Surgery. J Pediatr. 2015 Sep;167(3):599-604.e1-2. doi: 10.1016/j.jpeds.2015.06.035. Epub 2015 Jul 21. PMID 26205183
- [Background] Liu Y, Seipel C, Lopez ME, Nuchtern JG, Brandt ML, Fallon SC, Manyang PA, Tjia IM, Baijal RG, Watcha MF. A retrospective study of multimodal analgesic treatment after laparoscopic appendectomy in children. Paediatr Anaesth. 2013 Dec;23(12):1187-92. doi: 10.1111/pan.12271. Epub 2013 Sep 25. PMID 24112856
- [Background] Alkhoury F, Malvezzi L, Knight CG, Diana J, Pasaron R, Mora J, Aserlind A, Stylianos S, Burnweit C. Routine same-day discharge after acute or interval appendectomy in children: a prospective study. Arch Surg. 2012 May;147(5):443-6. doi: 10.1001/archsurg.2012.132. PMID 22785642
- [Background] Stessel B, Theunissen M, Fiddelers AA, Joosten EA, Kessels AG, Gramke HF, Marcus MA. Controlled-release oxycodone versus naproxen at home after ambulatory surgery: a randomized controlled trial. Curr Ther Res Clin Exp. 2014 Nov 28;76:120-5. doi: 10.1016/j.curtheres.2014.10.001. eCollection 2014 Dec. PMID 25516773